CLINICAL TRIAL: NCT01588730
Title: Dynamic and Static Splinting as a Treatment for Plantar Faciiopathy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Dynasplint Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dyna-PF 2011
Record Dates: First submitted 2011-07-14; First posted 2012-05-01 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-08

CONDITIONS: Plantar Fasciitis; Plantar Fasciopathy
Keywords: PF; Dynasplint; ADFD; AFD; Plantar Fasciitis; plantar Fasciopathy
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dynasplint (Experimental): Dynamic Splinting utilizes the protocols of Low-Load, Prolonged-Duration Stretch (LLPS) with calibrated, adjustable tension to increase the Total End Range Time (TERT) to reduce contracture. This unit is worn at night while sleeping (6-8 hours).
  Interventions: Device: Ankle Dorsiflexion Dynasplint
- Static Splint (Active Comparator): The control group will be treated with a static splint for a minimum of 6 4 hours each night while sleeping with the end goal of 6-8 hours.
  Interventions: Procedure: Commercially Available Static Night splint

INTERVENTIONS:
Device: Ankle Dorsiflexion Dynasplint — Dynamic Splinting utilizes the protocols of Low-Load, Prolonged-Duration Stretch (LLPS) with calibrated, adjustable tension to increase the Total End Range Time (TERT) to reduce contracture. This unit is worn at night while sleeping (6-8 hours) and, this does not affect activities of daily living
  Arms: Dynasplint
Procedure: Commercially Available Static Night splint — A commericially avilable static night splint will be worn for 4-6 hours during rest.
  Arms: Static Splint

SUMMARY:
The purpose of this study is to compare the Ankle Dorsiflexion Dynasplint System (DS) to static night splint for the reduction of pain from Plantar Fasciitis (Fasciopathy).

ELIGIBILITY:
Inclusion Criteria:

* All patients will have had a history of at least 3 consecutive months of plantar heel pain well-localized to the plantar fascia.
* All patients will have failed an initial treatment of non-weight bearing plantar and Achilles stretching.
* Diagnosis will be confirmed by physical examination by a single physician (JPF) with a typical point of maximum tenderness over the medial tubercle of the calcaneus

Exclusion Criteria:

* rheumatoid arthritis
* local infection
* pregnancy
* patients with tumors
* unresolved fractures
* severe peripheral vascular disease
* history of prior plantar fascia surgery
* history of plantar fascia rupture
* age <18 years
* recent ( within 6 weeks) steroid injection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-06; Primary Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
FFI score | 16 weeks
  The primary outcome measure will be difference between the pretreatment and two month cumulative Foot Function Index (PS-FFI) score

SECONDARY OUTCOMES:
Pain subscale and SROM questionnaire | 2, 4 and 12 months
  Secondary outcome measures will include two month, four month, and twelve month overall heel pain reduction measured by the responses to the following questionnaires:
  1. Pain subscale of the validated Foot Function Index (PS-FFI)
  2. A patient-relevant outcome measures (SROM) questionnaire that included generic and condition -specific outcome measures related to pain, function, and satisfaction with the treatment outcome.

CONTACTS AND LOCATIONS:
Overall Officials: John Furia, MD, Principal Investigator — SUN Orthopaedic Group Inc
Locations (1):
- SUN Orthopaedic Group Inc, Lewisburg, Pennsylvania, United States

REFERENCES:
- [Background] Batt ME, Tanji JL, Skattum N. Plantar fasciitis: a prospective randomized clinical trial of the tension night splint. Clin J Sport Med. 1996 Jul;6(3):158-62. PMID 8792046
- [Background] Berlet GC, Anderson RB, Davis H, Kiebzak GM. A prospective trial of night splinting in the treatment of recalcitrant plantar fasciitis: the Ankle Dorsiflexion Dynasplint. Orthopedics. 2002 Nov;25(11):1273-5. doi: 10.3928/0147-7447-20021101-20. PMID 12452346
- [Background] Furia JP, Rompe JD .Extracorporeal shock wave therapy in the treatment of chronic plantar fasciitis and Achilles tendinopathy.Curr Opin Orthop 2007;18:102-111
- [Background] Furia JP. The safety and efficacy of high energy extracorporeal shock wave therapy in active, moderately active, and sedentary patients with chronic plantar fasciitis. Orthopedics. 2005 Jul;28(7):685-92. doi: 10.3928/0147-7447-20050701-17. PMID 16119283
- [Background] Mizel MS, Marymont JV, Trepman E. Treatment of plantar fasciitis with a night splint and shoe modification consisting of a steel shank and anterior rocker bottom. Foot Ankle Int. 1996 Dec;17(12):732-5. doi: 10.1177/107110079601701203. PMID 8973894
- [Background] Powell M, Post WR, Keener J, Wearden S. Effective treatment of chronic plantar fasciitis with dorsiflexion night splints: a crossover prospective randomized outcome study. Foot Ankle Int. 1998 Jan;19(1):10-8. doi: 10.1177/107110079801900103. PMID 9462907
- [Background] Probe RA, Baca M, Adams R, Preece C. Night splint treatment for plantar fasciitis. A prospective randomized study. Clin Orthop Relat Res. 1999 Nov;(368):190-5. PMID 10613168
- [Background] Rompe JD, Cacchio A, Weil L Jr, Furia JP, Haist J, Reiners V, Schmitz C, Maffulli N. Plantar fascia-specific stretching versus radial shock-wave therapy as initial treatment of plantar fasciopathy. J Bone Joint Surg Am. 2010 Nov 3;92(15):2514-22. doi: 10.2106/JBJS.I.01651. PMID 21048171
- [Background] Sheridan L, Lopez A, Perez A, John MM, Willis FB, Shanmugam R. Plantar fasciopathy treated with dynamic splinting: a randomized controlled trial. J Am Podiatr Med Assoc. 2010 May-Jun;100(3):161-5. doi: 10.7547/1000161. PMID 20479445
- [Background] Wapner KL, Sharkey PF. The use of night splints for treatment of recalcitrant plantar fasciitis. Foot Ankle. 1991 Dec;12(3):135-7. doi: 10.1177/107110079101200301. PMID 1791004